CLINICAL TRIAL: NCT07176546
Title: TAVNEOS for Otolaryngologic Manifestations of Granulomatosis With Polyangiitis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Robert Spiera, MD (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Robert Spiera, MD, Principal Investigator, Hospital for Special Surgery, New York
Organization: Hospital for Special Surgery, New York (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-1580
Record Dates: First submitted 2025-08-18; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Granulomatosis With Polyangiitis; Wegener's; GPA
Keywords: Tavneos; avacopan; GPA; ENT
MeSH Terms: conditions — Granulomatosis with Polyangiitis | interventions — avacopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAVNEOS (Active Comparator): BID dose of 30 mg TAVNEOS
  Interventions: Drug: Avacopan
- Placebo (Placebo Comparator): BID dose of 30 mg TAVNEOS-matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avacopan — BID dose of 30 mg TAVNEOS (3-10mg capsules)
  Other Names: TAVNEOS
  Arms: TAVNEOS
Drug: Placebo — BID dose of 30mg TAVNEOS-matching placebo (3-10mg capsules)
  Arms: Placebo

SUMMARY:
This is a single center double-blind placebo-controlled study. Patients with GPA and active ears, nose, and throat (ENT) disease in at least two ENT domains, as defined after endoscopic visualization of the upper airway and audiometric evaluation, if applicable, by a single otolaryngologist using a validated GPA ENT disease activity score, will be eligible for inclusion. Patients will be treated with standard of care (SOC) treatment as determined by their treating rheumatologist. In addition to SOC, patients will be randomized to receive TAVNEOS 30mg BID or placebo. Patients will be followed for 52 weeks with standardized ENT assessment along with rheumatologic evaluation of overall disease activity with BVAS.

ELIGIBILITY:
Inclusion Criteria:

* GPA diagnosis defined by score of ≥5 on 2022 ACR/EULAR Classification Criteria for GPA
* Active GPA (both newly diagnosed and relapsing disease) in the ENT domain within 1 month prior to screening, where the active disease is defined as a score of ≥2 on a GPA ENT disease activity score (7 items scored as 1= present 0= absent) performed by direct endoscopic visualization of the upper airway and audiometric evaluation, if applicable, by a single expert otolaryngologist. Items included in the GPA ENT disease activity score are:

  * Bloody rhinorrhea (Daily blood stained nasal discharge)
  * Objective stridor (Stridor assessed by doctor)
  * Inflammation on nasal examination (Ulcers, granulation, friable mucosa on rigid nasal endoscopy. Excluding crusting)
  * Inflammation on flexible laryngoscopy (Ulcers, granulation, friable mucosa in the larynx)
  * Inflamed TM*/middle ear (Persistent inflammation or granulation tissue in tympanic membrane/middle ear)
  * Sudden sensorineural hearing loss (30db drop in 3 frequencies within 72 hours)
* Other ENT/upper airway manifestations of active GPA observed during structured ENT exam including but not limited to lacrimal gland dacryocystitis and endobronchial disease
* Age 18 and older
* Willing and able to comply with treatment and follow-up procedures
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
* Willing and able to provide written informed consent
* Adequate liver function as defined by AST or ALT <2x Upper Limit of Normal

Exclusion Criteria:

* Creatinine >4.0mg/dl or GFR <15 at baseline or dependence on dialysis
* Respiratory failure requiring mechanical ventilatory support or had experienced alveolar hemorrhage requiring invasive pulmonary ventilation support anticipated to last beyond the screening period of the study
* Previous treatment with TAVNEOS within 6 months of screening
* Inability to comply with study and/or follow-up procedures at investigator discretion.
* Intravenous glucocorticoids in the 4 weeks prior to screening except as premedication prior to infusion of rituximab
* Pregnant or breast-feeding
* Any other known multi-system autoimmune disease including eosinophilic granulomatosis with polyangiitis (Churg-Strauss), systemic lupus erythematosus, IgA vasculitis (Henoch-Schonlein), rheumatoid vasculitis, Sjogren's syndrome, anti-glomerular basement membrane disease, or cryoglobulinemic vasculitis
* Required dialysis or plasma exchange within 12 weeks prior to screening
* Have had a kidney transplant
* Any of the following within 12 weeks prior to screening: symptomatic congestive heart failure requiring prescription medication, unstable angina (unless successfully treated with stent or bypass surgery), clinically significant cardiac arrhythmia, myocardial infarction or stroke
* History or presence of any form of cancer within the 5 years prior to screening, with the exception of excised basal cell or squamous cell carcinoma of the skin, or carcinoma in situ such as cervical or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis
* Evidence of tuberculosis based on interferon gamma release assay (IGRA), tuberculin purified protein derivative (PPD) skin test, or chest radiography (X rays or CT scan) done at screening or within 6 weeks prior to screening
* HBV, HCV, or HIV viral screening test showing evidence of active or chronic viral infection done at screening or within 6 weeks prior to screening
* Received a live vaccine within 4 weeks prior to screening
* WBC count less than 3500/uL, or neutrophil count less than 1500/uL, or lymphocyte count less than 500/uL before start of dosing
* Evidence of hepatic disease: AST, ALT, alkaline phosphatase, or bilirubin >3 times the upper limit of normal before start of dosing
* Known hypersensitivity to avacopan or inactive ingredients of the TAVNEOS capsules
* Participated in any clinical study of an investigational product within 30 days prior to screening or within 5 half-lives after taking the last dose
* Participated previously in an TAVNEOS study
* Concurrent use of strong inducers of the CYP450 ie. carbamazepine, phenobarbital, phenytoin, rifampin, or St. John's wort
* Known hypersensitivity to avacopan or inactive ingredients of the avacopan capsules (including gelatin, polyethylene glycol, or Cremophor)
* History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the patient at unacceptable risk for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in ENT remission without relapse | Week 52
  The proportion of patients in ENT remission without relapse in each treatment group at week 52 with no glucocorticoid (GC) exposure 4 weeks prior to week 52, where ENT remission is defined as a score of 0 on GPA ENT disease activity score

SECONDARY OUTCOMES:
Mean ENT disease activity score | Week 52
  Comparison of mean ENT disease activity scores between treatment groups at week 52
Change in ENT disease activity score | Between week 26 and week 52
  Change in ENT GPA disease activity score between week 26 and week 52
Proportion of patients in ENT remission with BVAS 0 at week 52 and sustained remission | Week 52
  Proportion of patients in remission with BVAS 0 at week 52 and sustained remission from week 26 to week 52 with BVAS 0 and no glucocorticoids for 4 weeks prior to assessment
Cumulative steroid dose | Through study completion, an average of 60 weeks
Duration of steroid-free remission | Through study completion, an average of 60 weeks
Change in Vasculitis Damage Index (VDI) | Week 52
  Change in VDI in the ENT domain at week 52
Sino-nasal Outcome Test (SNOT-22) | Through study completion, an average of 60 weeks
  Scale 0-110 (Higher score equals worse outcome)
ANCA-Associated Vasculitis Patient-Reported Outcome (AAV-PRO) | Through study completion, an average of 60 weeks
  Scale 0-119 (Higher score equals worse outcome)
Number of surgical procedures in the ENT domain required | Through study completion, an average of 60 weeks
  Number of surgical procedures in the ENT domain required during the study period
Number of ENT flares | Through study completion, an average of 60 weeks
  Number of ENT flares as measured by the rise in GPA ENT DAS (defined by an increase of ≥1 point on the GPA ENT DAS)
Time to ENT relapse | Through study completion, an average of 60 weeks
Number of GPA flares | Through study completion, an average of 60 weeks
  Number of GPA flares as measured by Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS-WG)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York; Lindsay Lally, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Hackensack Meridian School of Medicine - Advanced Lung and Airway Center, Edison, New Jersey
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No